CLINICAL TRIAL: NCT07320976
Title: First-in-Human Study of a Novel Conformal Pulsed-Field Ablation Balloon Catheter for Pulmonary Vein Isolation in Paroxysmal Atrial Fibrillation
Brief Title: FIH of PFBalloon for PVI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Hanxiong Liu, Professor, The Third People's Hospital of Chengdu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFBalloon-FIH
Record Dates: First submitted 2025-12-08; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Paroxysmal atrial fibrillation; Pulsed field ablation; pulmonary vein isolation; first-in-human
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PFA for PVI (Experimental): The participates received PVI using a PFBalloon catheter with a novel waveform (Biphasic, Bipolar, 750 V) under general anesthesia. The balloon was inflated with 10:1 saline/contrast mix. Deployment-volume was adjusted to achieve a ball-shape, for performing wide antral catheter ablation (WACA), and a pear-shape, for ablating PV antra, ensuring optimal tissue contact with 8 applications per vein.
  Interventions: Device: PVI with a novel PFA catheter

INTERVENTIONS:
Device: PVI with a novel PFA catheter — PVI with a PFBalloon catheter with 8 applications per vein

SUMMARY:
The goal of this clinical trial is to assess the safety and effectiveness of a conformal pulsed field ablation (PFA) balloon catheter for pulmonary vein isolation (PVI) in patients with paroxysmal atrial fibrillation (AF). It will also explore the durable effectiveness of this novel catheter through post-ablation remapping.

The main questions it aims to answer are:

Does the conformal PFA balloon catheter achieve absence of periprocedural primary adverse events (primary safety endpoint)? Does the conformal PFA balloon catheter achieve acute PVI (primary effectiveness endpoint) and durable PVI at three months post-ablation (secondary effectiveness endpoint)?

This is a first-in-human, single-center trial that employs a novel PFA balloon catheter with a biphasic, bipolar 750 V waveform. The balloon is inflated with a 10:1 saline/contrast mixture, with deployment volume adjusted to form a sphere shape for wide-antral PV ablation or a pear shape for targeted ostial-junction ablation to ensure optimal tissue contact.

Participants will:

Undergo PVI using the novel conformal PFA balloon catheter; Be monitored for periprocedural primary adverse events to assess safety; Undergo remapping at three months post-ablation to assess durable PVI; Undergo follow-up visits scheduled for seven-days, 30-days, three-months, six-months, and 12-months post-procedure. Recurrence assessment includes: 1) routine 12-lead ECG examination during each visit and 2) 24-hour or seven-day Holter monitoring at six and 12 months.

DETAILED DESCRIPTION:
Background

Atrial fibrillation (AF) is the most prevalent sustained cardiac arrhythmia globally, with an estimated incidence of 1.5-2.0% in the general population. This condition markedly diminishes quality of life, elevates stroke risk fivefold, triples the incidence of congestive heart failure, and is associated with increased overall mortality. These adverse consequences primarily result from rapid, irregular ventricular rates and ineffective atrial contraction, which compromise cardiac output. The ensuing atrial dyssynchrony promotes blood stasis, elevating the risk of thrombus formation and subsequent ischemic stroke. Diagnosis is confirmed by electrocardiographic (ECG) documentation of chaotic atrial electrical activity.

First-line management typically involves pharmacotherapy targeting either ventricular rate control or rhythm control-the restoration and maintenance of sinus rhythm. However, antiarrhythmic drugs are limited by proarrhythmic potential, diminishing long-term efficacy, and possible increased mortality, especially in patients with ventricular dysfunction. Catheter ablation offers superior outcomes, including reduced AF recurrence, fewer cardiovascular hospitalizations, and decreased arrhythmia relapse. Current guidelines recommend ablation for symptomatic, drug-refractory paroxysmal AF, with pulmonary vein isolation (PVI) established as the foundational procedural strategy.

Conventional thermal ablation using radiofrequency or cryoenergy is an established, effective treatment for achieving PVI. However, the non-selective nature of thermal energy carries a risk of collateral damage to adjacent structures, potentially leading to rare but serious complications. Each modality presents specific trade-offs: radiofrequency ablation is technically demanding and time-intensive, while cryoballoon ablation offers ease of use but less precision for ablating non-pulmonary vein targets.

Pulsed field ablation (PFA) utilizes high-voltage, ultra-rapid electrical pulses to induce irreversible electroporation and non-thermal cell death. This energy source demonstrates high cardiomyocyte selectivity, thereby sparing adjacent critical structures such as the esophagus, phrenic nerve, and pulmonary veins. Notably, PFA has not been associated with typical thermal complications like atrioesophageal fistula, phrenic nerve palsy, or pulmonary vein stenosis. By minimizing collateral injury, PFA holds promise for enhancing the safety profile of PVI without compromising efficacy.

A novel, single-shot, 24-electrode, conformable balloon-based PFA catheter has been developed. Its design incorporates mid-voltage (750V) biphasic pulses delivered in a bipolar fashion between balloon electrodes, integrated tissue-contact verification, and conformability to accommodate variable anatomy. This report details the first-in-human experience evaluating this novel conformable PFA balloon catheter for PVI in patients with paroxysmal AF, assessing procedural performance, safety, acute effectiveness, and PVI durability via invasive remapping.

Methods

Study Design This prospective, single-arm, single-center, first-in-human (FIH) trial evaluated the safety and effectiveness of a novel conformable PFA balloon catheter (PFBalloon™, EnChannel Medical, China) for treating paroxysmal AF. The protocol was approved by the local Ethics Committee and conducted in accordance with the Declaration of Helsinki. All participants provided written informed consent. Enrolled subjects underwent first-time PVI and are being followed for 12 months post-ablation.

Study Population Eligible patients were aged 18-75 years with documented symptomatic paroxysmal AF (episode duration <7 days), who were refractory or intolerant to at least one Class I or III antiarrhythmic drug. Key exclusion criteria included reversible or non-cardiac causes of AF, prior AF ablation or surgery, anticipated need for extra-PVI ablation, persistent AF, left atrial diameter >50 mm, left ventricular ejection fraction <40%, presence of an implantable cardiac device, or intracardiac thrombus.

Procedural Workflow After enrollment and baseline bloodwork, left atrial computed tomography angiography was performed for thrombus exclusion and anatomical assessment. Pre-procedure, thrombus was further ruled out by transesophageal echocardiography. Phrenic nerve function was evaluated via diaphragmatic motion during inspiration and direct pacing before and after ablation.

Procedures were performed under general anesthesia. Following femoral venous access, intravenous heparin was administered to maintain an activated clotting time ≥300 seconds. Pre-ablation electroanatomic mapping was performed using a PENTARAY® catheter with the CARTO™ 3 system (Biosense Webster, USA).

The PFA balloon catheter was positioned in the left atrium over a guidewire. PVI was performed sequentially (left superior/inferior, then right superior/inferior veins). Each vein received eight PFA applications: four at the antrum with the balloon in a spherical configuration and four at the ostium with a pear-shaped configuration, achieved by adjusting contrast inflation volume. The catheter was slightly rotated after every two applications. Positioning was optimized using fluoroscopically-guided contrast injection. Conduction block was confirmed after a 20-minute waiting period, and post-ablation voltage mapping verified acute isolation. Additional lesions were applied if necessary.

Brain Magnetic Resonance Imaging Brain MRI with diffusion-weighted imaging was performed within 72 hours pre-procedure and 48 hours post-procedure to screen for acute silent cerebral ischemic events. Scans were reviewed by independent neuroradiologists.

Follow-up Post-ablation antiarrhythmic drug use was permitted per operator discretion and discontinued after three months. Oral anticoagulation was continued per guidelines. All patients underwent repeat invasive electrophysiological mapping at 90 days. Clinical follow-up occurred at 7 days, 30 days, 3, 6, and 12 months. Recurrence was assessed via 12-lead ECG at each visit and 24-hour or 7-day Holter monitoring at 6 and 12 months.

Study Endpoints The primary safety endpoint was the incidence of primary adverse events (PAEs) within 7 days post-ablation. Later-occurring events (device/procedure-related death, atrio-esophageal fistula, PV stenosis) were also considered PAEs. Persistent diaphragmatic paralysis/phrenic nerve palsy at 3 months were classified as PAEs.

The primary effectiveness endpoint was acute procedural success, defined as confirmation of entrance/exit block in all targeted pulmonary veins. Secondary effectiveness endpoints included: 1) patient-based durable PVI rate at 3-month remapping, 2) vein-based durable isolation rate at 3-month remapping, and 3) clinical efficacy at one year.

ELIGIBILITY:
1. Inclusion Criteria:

1. Aged 18-75 years
2. Documented symptomatic paroxysmal atrial fibrillation with episode duration <7 days
3. Refractory or intolerant to at least one Class I or III antiarrhythmic drug

2. Exclusion Criteria:

1. Atrial fibrillation caused by reversible or non-cardiac factors
2. Prior AF ablation or cardiac surgery history
3. Anticipated need for extra-pulmonary vein isolation (extra-PVI) ablation
4. Persistent atrial fibrillation
5. Left atrial diameter >50 mm
6. Left ventricular ejection fraction <40%
7. Presence of an implantable cardiac device (e.g., pacemaker, implantable cardioverter-defibrillator)
8. Intracardiac thrombus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Primary Adverse Events Within 3 Months Post-Ablation [Primary Safety Endpoint] | Within 3 months post-ablation.
  The primary safety endpoint was the incidence of primary adverse events (PAEs) within 7 days post-ablation. Later-occurring events (device/procedure-related death, atrio-esophageal fistula, PV stenosis) were also considered PAEs. Persistent diaphragmatic paralysis/phrenic nerve palsy at 3 months were classified as PAEs.
Acute Procedural Success: Confirmation of Entrance/Exit Block in All Targeted Pulmonary Veins [Primary Effectiveness Endpoint] | Immediately after the ablations
  The primary effectiveness endpoint was acute procedural success, defined as confirmation of entrance/exit block in all targeted pulmonary veins.

SECONDARY OUTCOMES:
Patient-Based Durable Pulmonary Vein Isolation (PVI) Rate at 3-Month Remapping [Secondary Effectiveness Endpoint] | 3 months post the index ablation procedure.
  The outcome measure is defined as the proportion of patients who maintain complete and durable isolation of all targeted pulmonary veins (without recurrence of conduction) at 3-month remapping after the index ablation procedure.
Vein-Based Durable Pulmonary Vein Isolation Rate at 3-Month Remapping [Secondary Effectiveness Endpoint] | 3 months post the index ablation procedure.
  The outcome measure is defined as the proportion of all targeted pulmonary veins that maintain complete and durable isolation (without recurrence of conduction) at 3-month remapping after the index ablation procedure.
1-Year Clinical Efficacy Assessed by Freedom from Atrial Fibrillation (AF) Recurrence [Secondary Effectiveness Endpoint] | 1 year post the index ablation procedure.
  The outcome measure is defined as the proportion of patients who remain free from recurrent atrial fibrillation (AF) (including symptomatic and asymptomatic AF, as confirmed by 12-lead electrocardiogram or 72-hour Holter monitoring) within 1 year after the index ablation procedure. Recurrence is defined as any episode of AF lasting ≥30 seconds after the 3-month blanking period.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third People's Hospital of Chengdu, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2-year sharing window post-publication
Access Criteria: 1. Eligible Recipients Qualified researchers with academic/institutional affiliation, who submit a feasible research proposal and agree to comply with data protection regulations.
  2. Access Process Submit application to the corresponding author via designated email.